CLINICAL TRIAL: NCT02671188
Title: A Multi-centre, Randomised, Double-blind (Sponsor Open), Placebo-controlled, Repeat Dose, Proof of Mechanism Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Efficacy of GSK3050002 in Subjects With Psoriatic Arthritis
Brief Title: A Study to Evaluate the Safety, Mode of Action and Clinical Efficacy of GSK3050002 in Subjects With Psoriatic Arthritis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was stopped before any subjects were treated, consequently there are no results for the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200928
Record Dates: First submitted 2016-01-18; First posted 2016-02-02 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Autoimmune Diseases
Keywords: C-C chemokine receptor; Psoriatic arthritis; Chemokine (C-C motif) ligand 20; Monoclonal antibody; psoriasis; Humanized Immunoglobulin G
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Psoriatic; Psoriasis | interventions — GSK3050002

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK3050002 100 mg/mL (Experimental): Subjects will be administered GSK3050002 intravenously (IV) over the period of approximately 2 hours on Day 1, Day 15 and Day 29 (total of 3 doses) in a clinical facility with regular monitoring of vital signs. Monitoring of vital signs will continue for a minimum of 2 hours after completion of Infusion. On Day 1, loading dose of GSK3050002 10 milligrams per kilogram (mg/kg) will be administered intravenously, followed by maintenance doses of 5mg/kg IV administered at Day 15 and Day 29. Each subject will receive a cumulative dose of 20 mg/kg.
  Interventions: Drug: GSK3050002
- Placebo (Placebo Comparator): Subjects will be administered normal saline (0.9% sodium chloride) intravenously over the period of approximately 2 hours on Day 1, Day 15 and Day 29 (total of 3 doses) in a clinical facility with regular monitoring of vital signs. Monitoring of vital signs will continue for a minimum of 2 hours after completion of Infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3050002 — The 3 mL glass vial contains white to off-white lyophilized powder which requires reconstitution with sterile water for injection.Prepared as 100 milligrams per milliliter (mg/mL) solution; lower concentrations prepared by dilution with 0.9% weight by volume (w/v) sodium chloride Injection for infusion.
  Arms: GSK3050002 100 mg/mL
Drug: Placebo — Normal saline (0.9% sodium chloride) will be used as placebo.
  Arms: Placebo

SUMMARY:
Chemokine (C-C motif) ligand 20 (CCL20) is a protein involved in attracting immune cells including subsets of T cells (for example Th17 cells), B cells, natural killer cells and dendritic cells to inflamed tissues in conditions such as psoriasis (Ps) and psoriatic arthritis (PsA). CCL20 acts by binding and activating the chemokine receptor 6 (CCR6) present on the surface of the inflammatory cells. Levels of CCL20 are increased in inflamed tissues in psoriasis (Ps) and inflammatory arthritis. GSK3050002 is a humanized Immunoglobulin G (Ig)G monoclonal antibody, which binds to and neutralizes the action of human CCL20. The hypothesis is that GSK3050002 will reduce the movement of inflammatory cells into tissues affected by Ps or PsA, thereby leading to an improvement in disease activity. The primary objective of this multi-centre, randomized, double-blind (sponsor open), placebo-controlled trial is to evaluate the safety and tolerability of repeat doses of GSK3050002, and to understand the mechanism of action (by taking skin and synovial biopsy samples) and potential for clinical efficacy of GSK3050002 in subjects with PsA. A minimum of 18 subjects and up to a maximum of 30 subjects will be randomised into the study to either GSK3050002 or placebo in a 2:1 ratio to ensure that approximately 18 evaluable subjects complete the study. The total duration of participation in the study will be approximately 21 weeks from screening to last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years and <=75 years of age at the time of consent.
* Diagnosis of, and currently active psoriatic arthritis with >=3 tender and >=3 swollen joints, one of which must be either a knee or ankle joint suitable for synovial biopsies.
* C-reactive protein (CRP) >=3mg/l at the time of screening, thought by the investigator to be due to active PsA.
* A negative test result for Rheumatoid Factor at screening.
* Active PsA despite an adequate course of treatment with at least one of the following Disease-modifying anti-rheumatic drugs (DMARDS): methotrexate, sulfasalazine or leflunomide for a minimum of 3 months, with a stable dose prior to screening. The subject may have received prior treatment for their PsA with up to three oral DMARDS.
* At least 2 active psoriatic skin lesions >=3centimetre (cm) x 3cm diameter at the time of the screening visit which in the opinion of the investigator will still be present in the Pre- Treatment Phase. Each plaque should have a total PLSS of >=5, including an induration score of >=2 (moderate or above) and a score of >=1 in erythema and scaling. The PLSS is the sum of the erythema, scaling and induration scores. The skin lesions should be located in areas usually shielded from natural light by clothing (e.g. trunk or proximal extremities) and should not include scalp, inguinal or genital lesions.
* BMI within the range 18 - 35 kilogram per squared meter (kg/m^2) (inclusive).
* Female subjects are eligible to participate if they are not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: 1. Pre-menopausal females with one of the following: a. Documented tubal ligation; b. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; c. Hysterectomy; d. Documented Bilateral Oophorectomy; e. Reproductive potential and agrees to follow one of the options listed below in the GSK (GlaxoSmithKline) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until 12 weeks after the last dose of study medication and completion of the follow-up visit at Day 113.

  2. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 12 weeks after the last dose of study medication:Vasectomy with documentation of azoospermia; Male condom plus female partner use of one of the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Childbearing potential listed below. GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penilevaginal intercourse on a long term and persistent basis. a. Contraceptive subdermal implant effectiveness criteria including a <1% rate of failure per year, as stated in the product label. b. Intrauterine device or intrauterine system that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label c. Oral Contraceptive, either combined or progestogen alone d. Injectable progestogen e. Contraceptive vaginal ring f. Percutaneous contraceptive patches g.Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.
* Capable of giving signed informed consent which includes compliance with study procedures and requirements as listed in the consent form and in this protocol

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Planned surgical joint procedure, including intra-articular, tendon sheath, or bursal corticosteroid injections, during the study.
* Intra-articular corticosteroid injection, arthrocentesis or synovial biopsy on the joint that has been identified for biopsy or Magnetic resonance imaging (MRI) within 6 weeks of the Pre-Treatment biopsy and MRI.
* Has undergone surgery, including synovectomy or arthroplasty, on the joint chosen for biopsy or MRI.
* History of joint disease, other than PsA, at the knee or ankle joint chosen for biopsy and/or MRI (eg gout, pseudogout, osteoarthritis).
* Diagnosed with a major chronic inflammatory or connective tissue disease other than Ps and PsA (e.g. rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, ankylosing spondylitis).
* An active infection, or a history of infections as follows: a. A serious infection, defined as requiring hospitalization or intravenous antiinfectives within 8 weeks prior to Day 1. b. Oral anti-microbials within 14 days of Day 1. c. A history of opportunistic infections within 1 year of screening (e.g. pneumocystis jirovecii, cytomegalovirus pnemonitis, aspergillosis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature d.Recurrent or chronic infection or other active infection that, in the opinion of the investigator might cause this study to be detrimental to the subject e. History of Tuberculosis (TB), irrespective of treatment status f. A positive diagnostic TB test at screening defined as a positive QuantiFERON®-TBGold (Registered product of QFT-G; Cellestis Ltd., Carnegie, Australia) test or T-spot test. In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative, or they have a negative Tuberculin Purified Protein Derivative (PPD) skin test. A positive PPD (Mantoux) test is defined as >=5mm of induration (size of raised lump not redness).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Known bleeding or coagulation disorder.
* Alanine aminotransferase (ALT) and bilirubin >1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QT interval corrected (QTc) > 450 milliseconds (msec), or QTc > 480 msec in subjects with Bundle Branch Block. If a single QTc is abnormal, then the averaged QTc values of triplicate ECGs obtained (each separated by at least 5 min) will be utilized to determine eligibility.
* Active malignancy or carcinoma in situ in the past 5 years. There is an exception for basal cell carcinoma or cervical carcinoma in situ if they have had curative surgical treatment.
* Significant unstable acute illness or uncontrolled chronic disease other than PsA, which in the opinion of the investigator, would preclude the subject from study participation.
* Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but not limited to: a. Intracranial aneurysm clips (except Sugita) or other metallic objects, b. History of intra-orbital metal fragments that have not been removed by a medical professional, c.Pacemakers or other implanted cardiac rhythm management devices and non-MR compatible heart valves, d.Inner ear implants, e.History of claustrophobia which may impact participation.
* Receiving treatment with anti-coagulant medications, including warfarin, heparin, thrombin inhibitors, and Factor Xa inhibitors, unless the subject is able to discontinue these medications one week prior to biopsies in the Pre-Treatment Phase and at one week prior to the Day 43 biopsies, unless local guidelines indicate a different timeframe, in which case local guidelines may be followed, taking into account the risk:benefit and the indication for use of those medications. The anticoagulants may be re-started 3 days after the biopsy, or according to local guidelines.
* Received treatment with the therapies listed below, within the prescribed timeframe. If in doubt, or the therapy is not listed, please consult with the medical monitor. Treatment with, cyclosporine, tacrolimus, hydroxychloroquine, azathioprine (28 days prior to Screening until Follow-up) apremilast or tofacitanib (At any time prior to Screening until Follow-up). Intravenous, intra-muscular or intra-articular glucocorticoids (28 days prior to screening until follow up). Topical psoriasis therapies (other than on face and genitals where topical therapy may continue during the study) (14 days prior to Screening until Follow-up).Emollients are allowed except on the day of study visits prior to assessments. Biologic therapies for the treatment of psoriasis, psoriatic arthritis or inflammatory arthritis including but not limited to anti-tumor necrosis factors biologics, etanercept, ustekinumab, secukinumab, rituximab, abatacept or tocilizumab (At any time prior to Screening until Follow-up). Alkylating agents (chlorambucil, cyclophosphamide) (At any time prior to Screening until Follow-up) Investigational biological and nonbiological immunomodulatory therapies (At any time prior to Screening until Follow-up). Psoralen long wave ultraviolet radiation treatment (28 days prior to Screening until Follow-up) Acitretin/Retinoids (28 days prior to Screening until Follow-up). Single treatment phototherapy (Ultraviolet B or self therapy with tanning bed or solarium) (14 days prior to Screening until Follow-up). Live vaccination Live vaccinations are not permitted within (28 days of first dose until 12 weeks after the last dose). If indicated, non-live vaccines (e.g. inactivated influenza vaccines) may be administered whilst receiving GSK3050002 based on an assessment of the benefit: risk (e.g. risk of Therapy Time period decreased responsiveness). Investigators are expected to follow local and/or national guidelines with respect to vaccinations, including against influenza and pneumococcus, in subjects with PsA.
* A history of drug and alcohol misuse that could interfere with participation in the trial according to the protocol, or in the opinion of the investigator impacts on the physical or mental wellbeing of the subject.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation. This include a history of severe drug allergies, including Type I hypersensitivity reactions to parenteral administration of human or murine proteins or monoclonal antibodies.
* Contraindication to gadolinium contrast agent in accordance with local guidelines.
* Presence of hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Platelet count is <100 x 10^9/mL or prothrombin time is above the laboratory upper limit of normal at screening.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Estimated GFR (Modification of Diet in Renal Disease [MDRD] calculation) of less than 60 milliliters per minute (mL/min) per 1.73 squared meter /m^2 at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-08-09 (Estimated); Study Completion 2019-08-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AE) | Up to Day 116
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of subjects with Serious Adverse Events | Up to Day 116
  An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the subjects or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, and is associated with drug-induced liver injury.
Composite of clinical laboratory assessments as a measure of safety and tolerability. | Up to Day 116
  Clinical laboratory assessments will include hematology, clinical chemistry and urinalysis.
Composite of vital signs as a measure of safety and tolerability. | Up to Day 116
  Vital signs to be measured in semi-supine position after at least 5 minutes rest and will include temperature, systolic and diastolic blood pressure, and pulse rate.
Electrocardiogram (ECG) assessment as a measure of safety and tolerability. | Up to Day 116
  A single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and corrected QT (QTc) intervals.

SECONDARY OUTCOMES:
GSK3050002- CCL20 complex levels in serum | Baseline and Up to Day 116
  Blood samples will be collected on baseline (Day-10 to -1), at pre-dose and at 120 minutes post start of infusion, immediately after infusion has ceased on D 15 and D 29, D 43, D 85, D 113 +/- 3 days
Change from baseline in the number of CD3+ T cells synovial tissue and skin biopsy in samples | Baseline and Day 43
  Synovial and skin lesion biopsy tissue will be collected and evaluated for general appearance and inflammatory infiltrate including CD3+ T-cells
Change from baseline in Disease Activity Score 28 (DAS28) | Baseline and Up to Day 116
  DAS28 is a composite arthritis disease activity index comprising swollen and tender joint count (28 joints), patient global assessment of disease activity, and C-reactive protein.
Changes in American College of Rheumatology (ACR) responders | Baseline and Up to Day 116
  ACR is a composite score of the patient assessment of joint pain, the patient global assessment of disease activity, the physician global assessment of disease activity, the 66/68 swollen/tender joint count, the Disability Index of the Health Assessment Questionnaire (HAQ-DI) questionnaire, and C-reactive protein. The ACR is reported as % improvement (20%, 50% or 70%), between two discrete timepoints, as calculated by improvement in the 66/68 swollen/tender joint count, and improvement in at least three of the remaining five composite parameters.
Changes from baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) | Baseline and Up to Day 116
  PASDAS is a composite disease activity index for psoriatic arthropathies comprising the 66/68 swollen/tender joint count, patient global assessment of disease activity, physician global assesment of disease activity, Leeds enthesitis index, dactylitis score, SF-36 questionnaire and C-reactive protein
Changes in Psoriasis Lesion Severity Score (PLSS) | Baseline and Up to Day 116
  The PLSS is the sum of the erythema, scaling and plaque thickness scores.
Changes in Psoriasis Area Severity Index (PASI) | Baseline and Up to Day 116
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), thickness (induration), and scale, as well as the extent of body surface area (BSA) affected with psoriasis. Higher scores indicate more severe disease. PASI is a static measurement made without reference to previous scores
Incidences of serum anti- GSK3050002 antibody levels | Baseline and Up to Day 116
  Serum samples will be collected from all subjects at pre-dose and various time points post-dosing. An assay for detecting Anti-drug Antibodies (ADAs) against GSK3050002 will be done using validated electrochemiluminescent (ECL) bridging assay and the Meso-Scale Discovery (MSD) technology.
Titres of serum anti- GSK3050002 antibody levels | Baseline and Up to Day 116
  The serum which contain potential anti-GSK3050002 antibodies will be confirmed by immunocompetition using excess drug. Confirmed samples with ADA will be further analyzed for titers.
Maximum serum concentrations (Cmax) after repeat dosing of GSK3050002 | Up to Day 116
  Blood samples were collected at pre-dose and at 120 minutes post start of infusion, immediately after infusion has ceased on Day (D)1, D15, and D29. Blood samples were also collected D 8, D 22, D 43, D 57, D 85 and D 113 +/-3 days.
Area under curve over the dosing interval AUC (0- tau) after repeat dosing of GSK3050002 | Up to Day 116
  Blood samples were collected at pre-dose and at 120 minutes post start of infusion, immediately after infusion has ceased on Day (D)1, D15, and D29. Blood samples were also collected D 8, D 22, D 43, D 57, D 85 and D 113 +/-3 days.
Systemic clearance (CL) after repeat dosing of GSK3050002 | Up to Day 116
  Blood samples were collected at pre-dose and at 120 minutes post start of infusion, immediately after infusion has ceased on Day (D)1, D15, and D29. Blood samples were also collected D 8, D 22, D 43, D 57, D 85 and D 113 +/-3 days.
Volume of distribution (V) after repeat dosing of GSK3050002 | Up to Day 116
  Blood samples were collected at pre-dose and at 120 minutes post start of infusion, immediately after infusion has ceased on Day (D)1, D15, and D29. Blood samples were also collected D 8, D 22, D 43, D 57, D 85 and D 113 +/-3 days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Oxford, United Kingdom